CLINICAL TRIAL: NCT05750875
Title: Comparison of the Efficacy of Gabapentin With Loratadine in the Treatment of Uremic Pruritus in Patients of Chronic Kidney Disease
Brief Title: Gabapentin Versus Loratadine in Uremic Pruritus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Fawad Ahmad Randhawa, Associate Professor of Endocrinology, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9669/REG/KEMU/2021
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Pruritus; Uremia; Chronic Kidney Diseases
Keywords: Efficacy; Gabapentin; Loratadine; Uremic Pruritus
MeSH Terms: conditions — Pruritus; Uremia; Renal Insufficiency, Chronic | interventions — Loratadine; Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Loratadine (Active Comparator)
  Interventions: Drug: Loratadine
- Gabapentin (Active Comparator)
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Loratadine — Participants were given loratadine 10mg, oral, daily, for 4 weeks
  Arms: Loratadine
Drug: Gabapentin — Participants were given gabapentin 100mg, oral, daily, for 4 weeks
  Arms: Gabapentin

SUMMARY:
The goal of this clinical trial is to compare the efficacy of gabapentin with loratadine in reducing the severity of uremic pruritus in patients of chronic kidney disease and to compare the side effects of both drugs. The main questions it aims to answer are:

* Which drug (gabapentin versus loratadine) is more effective in reducing the severity of uremic pruritus?
* Which drug (gabapentin versus loratadine) has fewer side effects?

Participants were divided into two groups.Group A received loratadine 10mg daily and group B received gabapentin 100mg daily. Both groups were given treatment for 4 weeks.

* Participants were asked to grade the severity of pruritus on a numerical rating scale and also answer the Dermatology Life Quality Index Questionnaire (DLQI)
* Participants were also asked to report any side effects, if occurred.

Researchers compared both groups with regards to improvement in pruritus severity, DLQI score and side effects.

DETAILED DESCRIPTION:
Informed written consent was taken from all the participants. Participants were asked to discontinue any topical or systemic antipruritic drugs, for least 1 week prior to the study. Demographic, clinical and laboratory data (complete blood count, renal function tests, liver function tests, serum electrolytes and ultrasound abdomen) was evaluated at baseline. Glomerular Filtration Rate (GFR) and stage of chronic kidney disease was calculated. Participants were randomly allocated to two groups. One group received loratadine 10mg daily and the other received gabapentin 100mg daily. Those participants undergoing hemodialysis received their respective dose after the dialysis session. Both groups were given treatment for 4 weeks. Participants were asked to grade the severity of pruritus on a numerical rating scale and also answer the Dermatology Life Quality Index Questionnaire.These proformas were filled once at the start of the study, at 2 weeks and then at the end of study i.e. 4 weeks. Participants were also asked to report any adverse events, if occurred.

The Statistical Package for the Social Sciences (SPSS) version 25.0 was used to analyze the data. Qualitative data (like gender, dialysis status, etc.) was expressed in the form of frequency and percentages while quantitative data (like age, weight, serum creatinine levels, etc.) was represented as mean and standard deviations (Mean±SD). The reduction in scores of numerical rating scale and Dermatology Life Quality Index Questionnaire was calculated from baseline. Mean reduction in scores were compared between the two groups and independent sample t-test was applied. p-value <0.05 was considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease, stage 3 and above, irrespective of dialysis status
* Persistent pruritus, of moderate to very severe intensity (≥ 4 points on numerical rating scale), occurring at least 3 times a week, for at least 2 weeks, in a 1-month period.

Exclusion Criteria:

* Chronic skin conditions such as eczema, psoriasis, etc.
* Pruritus due to any other cause, such as metabolic abnormalities, liver disease, etc.
* History of drugs causing pruritus such as opioids, etc
* Pregnant patients
* Preceding history of allergy to either gabapentin or loratadine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Mean reduction in pruritus score, from baseline till 4 weeks, as measured on a numerical rating scale. | Four weeks
  Reduction in pruritus score as measured on a numerical rating scale, numbered between '0' (corresponding to no itch) and '10' (the worst imaginable itch).

SECONDARY OUTCOMES:
Mean reduction in Dermatology Life Quality Index Questionnaire score, from baseline till 4 weeks. | Four weeks
  Dermatology Life Quality Index Questionnaire score ranging from from 0 (no impairment of life quality) to 30 (maximum impairment).
Comparison of side effects of gabapentin and loratadine, as reported by the participants. | Four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Noor-Un-Nisaa Zia, MD Medicine, Principal Investigator — King Edward Medical University
Locations (1):
- King Edward Medical University/Mayo Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT05750875/Prot_ICF_000.pdf